CLINICAL TRIAL: NCT00005379
Title: Tuberculosis in a Multiethnic Inner City Population
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 4283; R01HL051517 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2015-12-29 (Estimated); Status verified 2015-12

CONDITIONS: Acquired Immunodeficiency Syndrome; HIV Infections; Lung Diseases; Tuberculosis; Mycobacterium Tuberculosis
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; HIV Infections; Lung Diseases; Tuberculosis

STUDY DESIGN:
Observational Model: Case-Control

GROUPS / COHORTS (3):
- IV drug users and their sexual contacts: This group will be made up of an already-recruited cohort
- Children who receive primary care at Bellevue Hospital
- Bellevue Hospital inpatients/outpatients: Inpatients being treated for TB and outpatients receiving prophylactic treatment

SUMMARY:
To determine the incidence of tuberculosis in an inner city population, identify risk factors for TB, describe the natural history in adults and children, evaluate the effect of Mycobacterium tuberculosis (Mtb) co-infection on the progression of human immunodeficiency virus disease, and determine factors that contribute to compliance and non-compliance with prophylaxis and treatment.

DETAILED DESCRIPTION:
BACKGROUND:

The research provided urgently needed information regarding incidence, risk factors, natural history, molecular epidemiology, treatment, and prevention of tuberculosis in an especially vulnerable multi-ethnic inner-city population with a high HIV seropositivity rate.

The study was part of a collaborative project on minority health, The Epidemiology, Drug Resistance, and Therapy of Tuberculosis in a Multi-Ethnic Inner City Population with a High HIV Seropositivity Rate. The 1993 Report of the Committee on Appropriations, House of Representatives, encouraged the NHLBI to establish minority centers to facilitate the diagnosis and treatment of cardiovascular diseases. The concept for the initiative was developed by the NHLBI staff and approved by the September 1992 National Heart, Lung, and Blood Advisory Council. The Request for Applications was released in October 1992.

DESIGN NARRATIVE:

The study was conducted prospectively and retrospectively in three groups of patients: intravenous drug users and their sexual contacts in an already-recruited cohort; children who received their primary care at Bellevue Hospital Medical Center; and Bellevue Hospital Center inpatients with TB and outpatients who underwent prophylactic treatment. In addition to environmental risk factors (e.g., hopelessness, cohabitation with tuberculosis patients and injected drug use), host factors were investigated, including: HIV infection; immune status among HIV- seropositive persons, as indicated by quantitative p24 antibodies; CD4, CD8, and gammadelta T cell counts; and race, age, and nutritional status. Incidence and risk-factors in the cohort were assessed by interview, blood draw, PPD screening, medical record review, and anergy panel. Natural history and impact on HIV disease in adult and pediatric populations were assessed by interviews, clinical screening and laboratory measures. Drug sensitivity testing and RFLP typing of specimens from the two populations were conducted, respectively, at the Bellevue Mycobacteriology Lab and the Public Health Research Institute. Factors affecting treatment compliance were assessed by self-administered questionnaire.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will be made up of three cohorts: (1) intravenous drug users and their sexual contacts in an already-recruited cohort; (2) children who receive their primary care at Bellevue Hospital Medical Center; and (3) Bellevue Hospital Center inpatients with TB and outpatients undergoing prophylactic treatment
Sampling Method: Non-Probability Sample
Dates: Start 1994-08; Primary Completion 1999-07 (Actual); Study Completion 1999-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Marmor, Principal Investigator — NYU Langone Medical Center

REFERENCES:
- [Background] Wolfe H, Marmor M, Maslansky R, Nichols S, Simberkoff M, Des Jarlais D, Moss A. Tuberculosis knowledge among New York City injection drug users. Am J Public Health. 1995 Jul;85(7):985-8. doi: 10.2105/ajph.85.7.985. PMID 7604926
- [Background] Davidow AL, Marmor M, Alcabes P. Geographic diversity in tuberculosis trends and directly observed therapy, New York City, 1991 to 1994. Am J Respir Crit Care Med. 1997 Nov;156(5):1495-500. doi: 10.1164/ajrccm.156.5.96-12078. PMID 9372666
- [Background] Davidow AL, Alcabes P, Marmor M. The contribution of recently acquired Mycobacterium tuberculosis infection to the New York City tuberculosis epidemic, 1989-1993. Epidemiology. 2000 Jul;11(4):394-401. doi: 10.1097/00001648-200007000-00006. PMID 10874545